CLINICAL TRIAL: NCT00973986
Title: Study the Effect of CYP3A Genetic Polymorphisms on the Pharmacokinetics of Atorvastatin in Chinese Subjects With Coronary Heart Disease
Brief Title: Effect of CYP3A Genetic Polymorphisms on the Pharmacokinetics of Atorvastatin
Acronym: ECGPPA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Liuhuaqiao Hospital (Other)
Collaborators: Guangdong Province, Department of Science and Technology (Other Government)
Responsible Party: Department of pharmacy, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YWLCSY-0900328; 08110831; GZJQZYY-003; ATR-01; GD080625; 20081001
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2009-09

CONDITIONS: Coronary Heart Disease
Keywords: atorvastatin; genetic polymorphisms; coronary heart disease; pharmacokinetics; CYP3A
MeSH Terms: conditions — Coronary Disease | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CYP3A4*1/*1 (Active Comparator)
  Interventions: Drug: Atorvastatin
- CYP3A4*1/*1G (Active Comparator)
  Interventions: Drug: Atorvastatin
- CYP3A4*1G/*1G (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — The subjects will receive atorvastatin (20 mg single dose) orally with approximately 240 ml of water. Blood samples(4 mL) will be taken prior to dosing and at 0.33, 0.66, 1, 1.5, 2, 2.5, 3, 4, 6, 9, 12, 24 and 48 h after drug administration.
  Other Names: Lipitor; Atorvastatin Calcium Tablets

SUMMARY:
The aim of the study is to investigate the effects of CYP3A polymorphisms on the pharmacokinetics of Atorvastatin in Chinese subjects with coronary heart disease.

DETAILED DESCRIPTION:
Large variability exists in the individual response to statins. CYP3A polymorphisms likely contribute to variable response to those drugs primarily metabolized by CYP3A including atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subjects must be >=35 years and <=70 years of age.
* Subjects must have an LDL-C concentration >=2.6 mmol/L and TC concentration >=4.14 mmol/L
* Body mass index (BMI) must be within the range of 19 to 30 for patients.
* Subjects must have documented coronary heart disease with one or more of the following features:

  * Documented stable angina (with evidence of ischemia on exercise testing)
  * History of myocardial infarction
  * History of percutaneous coronary intervention (with or without stent placement)
  * Documented history of unstable angina or non-Q wave myocardial infarction.

Exclusion Criteria:

* Diabetes and endocrine or metabolic disease.
* Congestive heart failure defined by New York Heart Association (NYHA) as Class III or IV.
* Uncontrolled cardiac arrhythmia.
* Uncontrolled hypertension (Systolic BP >160 mm Hg and/or Diastolic BP >100 mmHg on two consecutive measurements).
* Liver or kidney disease confirmed by abnormal lab values or function.
* Smokers who report cigarette use of more then 10 cigarette per day.
* Subjects who consume >2 alcoholic drinks a day. (A drink is: a can of beer, glass of wine, or single measure of spirits).
* Known human immunodeficiency virus (HIV) positive.
* Cancer.
* Subjects who are on any of the following concomitant medications:

  * Medications that are potent inhibitors of CYP3A, including cyclosporine, itraconazole, fluconazole, and ketoconazole, erythromycin or clarithromycin, nefazodone, protease inhibitors,mibefradil and large amounts of grapefruit juice (>1 quart/day).
  * Lipid-lowering agent: niacin (>200 mg/day) taken within 5 weeks, fibric acid derivatives taken within 8 weeks.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Compare the area under the plasma concentration versus time curve (AUC) and Area under the plasma concentration versus time curve (AUC) of atorvastatin with different CYP3A4*1G genotypes. | 48h

SECONDARY OUTCOMES:
The pharmacokinetics of atorvastatin in Chinese with coronary heart disease. | 48h

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Shujin, PhD, Study Director — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] He BX, Shi L, Qiu J, Zeng XH, Zhao SJ. The effect of CYP3A4*1G allele on the pharmacokinetics of atorvastatin in Chinese Han patients with coronary heart disease. J Clin Pharmacol. 2014 Apr;54(4):462-7. doi: 10.1002/jcph.229. Epub 2013 Nov 27. PMID 24214373